CLINICAL TRIAL: NCT03176472
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of Ricolinostat in Patients With Painful Diabetic Peripheral Neuropathy
Brief Title: Ricolinostat in Patients With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regenacy Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REGY-DN-201
Record Dates: First submitted 2017-05-18; First posted 2017-06-05 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Painful Diabetic Peripheral Neuropathy
Keywords: Diabetic Neuropathic Pain; Neuropathic Pain; HDAC6; ricolinostat; Painful Diabetic Peripheral Neuropathy; DPN
MeSH Terms: conditions — Neuralgia | interventions — ricolinostat

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ricolinostat (Experimental): Ricolinostat 120 mg, taken once daily (QD) by mouth; each dose in 12 mL liquid formulation (10 mg ricolinostat per mL)
  Interventions: Drug: ricolinostat
- placebo (Placebo Comparator): Placebo, 12 mL of liquid formulation with no active ingredient (i.e., ricolinostat), taken once daily (QD) by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ricolinostat — 120 mg per dose in 12 mL liquid formulation
  Other Names: ACY-1215
  Arms: ricolinostat
Drug: Placebo — 12 mL liquid formulation placebo
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, 2-arm, parallel group study of up to 274 evaluable patients designed to evaluate the safety and efficacy of the histone deacetylase 6 (HDAC6) inhibitor ricolinostat for painful DPN.

DETAILED DESCRIPTION:
The study includes an approximately 12 week randomized, double-blind, placebo controlled Treatment period in which patients will receive either ricolinostat or placebo, followed by an approximately 12 week open label Safety Extension period during which all patients will receive ricolinostat 120 mg daily.

Prior to randomization, patients will be enrolled in a baseline Pain Observation period from Day -14 to Day -1, during which the NRS (average and worst pain) will be recorded daily using an electronic daily diary that will be completed by patients to allow patients to familiarize themselves with the pain rating procedures, and to establish a baseline and confirm eligibility to participate. Patients will also initiate daily dosing during this time to evaluate compliance eligibility for participation. A daily diary will be used by the patient to record the pain assessments and rescue medication use. A follow-up phone contact will be conducted at Day -7 to Day -5 to review diary and dosing compliance.

Following the baseline Pain Observation period, patients who meet entry criteria will be randomized in a 1:1 ratio to receive either ricolinostat or placebo. During the 12-week double-blind, placebo-controlled Treatment period, patients will return for assessments in accordance with the schedule of assessments. At the conclusion of the approximately 12 week open label Safety Extension period, patients will enter a Follow-up safety washout and assessment period, which will incorporate 2 visits at approximately 2 and 4 weeks following the final Safety Extension visit, with assessments performed as outlined in the schedule of assessments.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes of at least 6 months with optimized and stable glycemic control during the 3 months prior to Screening
* Painful distal symmetric sensorimotor polyneuropathy due to diabetes
* Douleur Neuropathique 4 (DN4) score of ≥4
* Satisfactory diary data during the 14-day Pain Observation period determined by an algorithm that includes diary compliance, overall level of pain and day-to-day variability in pain

Exclusion Criteria:

* Pregnant or lactating
* Body Mass Index (BMI) >40 kg/m2
* Presence of any neuropathy other than DPN and/or significant risk factors for neuropathy other than diabetes
* Other pain conditions that could confound the results of this study, or other chronic pain condition(s) that could affect compliance with pain medication restrictions or confound pain assessments
* Painful DPN patients who have undergone lower limb amputations, are non-ambulatory, or whose walking is so impaired as to require a walker or other assistance for ambulation
* Have met Diagnostic and Statistical Manual of Mental Disorders V (DSM V) criteria for opioid use disorder or alcohol use disorder
* Opioid use at a dose of ≥ 30 morphine milligram equivalents on 3 or more days a week during the month prior to Screening
* Suicidal ideation/behavior as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* The use of marijuana or cannabidiol (CBD) during the 30 days prior to starting study drug
* Chronic use of over-the-counter capsaicin on extremities within 3 months of Screening and/or prescription Qutenza use within 6 months of Screening
* Corrected QT interval at Screening using QTcF of ≥450 msec (male) or ≥460 msec (female)
* Hemoglobin < 11.5 g/dL (female) or < 13 g/dL (male), total white blood cell count < 2500/mm3, neutrophil count < 1250/mm3, lymphocyte count < 1000/mm3, or platelet count < 100,000/mm3
* HIV positive and/or active hepatitis virus (A, B, or C) infection
* Current or previous (≤1 month of Screening) enrollment in a clinical trial involving treatment with an investigational product
* Any known recent exposure within the 14 days prior to initial Screening to coronavirus disease 2019 (COVID-19) or symptoms of COVID-19 infection or other reason to suspect COVID-19 infection as assessed by the Investigator at the time of initial Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Diabetes/Lipid Management & Research Center, Huntington Beach, California
  - National Research Institute, Huntington Park, California
  - Altman Clinical and Translational Research Institute, La Jolla, California
  - Torrance Clinical Research Institute Inc, Lomita, California
  - Providence Clinical Research, North Hollywood, California
  - Center for Clinical Research Inc, San Francisco, California
  - Diablo Clinical Research Inc, Walnut Creek, California
  - Innovative Research of West Florida Inc, Clearwater, Florida
  - DeLand Clinical Research Unit, Lake Mary, Florida
  - ClinCloud LLC, Maitland, Florida
  - APF Research LLC, Miami, Florida
  - International Research Associates LLC, Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Research, Tampa, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - NY Scientific, Brooklyn, New York
  - Triad Clinical Trials, Greensboro, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Wasatch Clinical Research LLC, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Double Blind Treatment Period
Arm/Group | Ricolinostat | Placebo
Started | 142 | 140
Completed | 132 | 124
Not Completed | 10 | 16
Not completed — Withdrawal by Subject | 5 | 10
Not completed — Adverse Event | 0 | 5
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Not Provided | 1 | 0
Period: Open Label Extension
Arm/Group | Ricolinostat | Placebo
Started | 131 | 121
Completed | 123 | 109
Not Completed | 8 | 12
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Not Provided | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Intent To Treat (ITT) Population is defined as all randomized subjects regardless of study drug administration
Groups:
- Total: Total of all reporting groups
Arm/Group | Ricolinostat | Placebo | Total
Number analyzed (Participants) | 142 | 140 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.64) | 60.9 (7.81) | 60.2 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 83 | 169
  Male | 56 | 57 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 37 | 39 | 76
  White | 93 | 95 | 188
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Height [Mean (Standard Deviation); unit: centimeters] | 172.7 (9.82) | 173.1 (9.91) | 172.9 (9.85)
Weight [Mean (Standard Deviation); unit: Kg] | 93.7 (18.29) | 96.76 (16.50) | 95.22 (17.46)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.31 (4.91) | 32.21 (4.17) | 31.75 (4.57)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Average Pain Intensity (NRS)
Description: Difference between mean average pain intensity using the 11-point numerical pain rating scale (NRS) consisting of pain measurement from 0-10 with 10 being the worst pain and 0 being no pain at all.
Time Frame: Baseline week [Day-7 to Day 1] compared to Final week [12 Weeks]
Population: The number of subjects with non-missing values at both Baseline and specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ricolinostat | Placebo
Number analyzed (Participants) | 140 | 142
units on a scale | -1.21 (1.4) | -1.03 (1.4)

2. Secondary Outcome: Change in Non-pain Neuropathic Signs (UENS)
Description: Change in non-pain neuropathic signs utilizing the Utah Early Neuropathy Score (UENS) which is a physical examination-based scale designed to assess early sensory predominant polyneuropathy. Compared with other scales, the UENS emphasizes severity and spatial distribution of pin (sharp) sensation loss in the foot and leg and focuses less on motor weakness. The UENS utilizes a numeric scale from 0-42, with higher scores indicating greater disease severity.
Time Frame: Baseline week [Day-7 to Day 1] compared to Week 12
Population: The number of subjects with non-missing values at both Baseline and specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ricolinostat | Placebo
Number analyzed (Participants) | 141 | 139
units on a scale | -1.51 (0.39) | -1.84 (0.40)

ADVERSE EVENTS:
Time Frame: Baseline through 24 weeks
Groups:
- Open Label Extension: Ricolinostat 120 mg, taken once daily (QD) by mouth; each dose in 12 mL liquid formulation (10 mg ricolinostat per mL)
  ricolinostat: 120 mg per dose in 12 mL liquid formulation
Arm/Group | Ricolinostat | Placebo | Open Label Extension
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/140 | 0/252
Serious Adverse Events (participants affected / at risk) | 6/142 | 2/140 | 4/252
Other Adverse Events (participants affected / at risk) | 17/142 | 21/140 | 20/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ricolinostat (N=142) | Placebo (N=140) | Open Label Extension (N=252)
Complex Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Worsening diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
WORSENING CHRONIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Proximal RCA Stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
NASAL BONE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN, NON-CARDIAC (General disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
EPILEPTIC SEIZURES (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC ARREST EPISODES (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
SEVERE SYMPTOMATIC ORTHOSTATIC SEVERE HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
UNCONTROLED DIABETES (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
RIGHT FOOT CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PROXIMAL LAD STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
LIVER LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LEFT KNEE WOUND CONTAMINATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
BILATERAL UPPER EXTREMITIES RECOVERED/RESOLVED ABRASIONS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RIGHT FLANK ABRASIONS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LEFT KNEE LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TONGUE LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
BILATERAL LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SURGICAL SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ricolinostat (N=142) | Placebo (N=140) | Open Label Extension (N=252)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2)
Difficulty Swallowing (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Common Cold (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Facial Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocytic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03176472/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT03176472/SAP_001.pdf